CLINICAL TRIAL: NCT01621152
Title: Electronic Surveillance Sniffer for Early Detection and Intervention for Acute Kidney Injury: PRAISE Trial
Brief Title: PRevention of Acute Kidney Injury Initiated With Electronic Surveillance Enhancement
Acronym: PRAISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kianoush B. Kashani, Consultant in Nephrology and Critical Care Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 11-000007
Record Dates: First submitted 2012-05-14; First posted 2012-06-18 (Estimated); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Acute Kidney Injury
Keywords: Acute renal failure; acute kidney injury; electronic surveillance; AKI; sniffer; AKIN; improvement in the process of care and outcomes
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional management arm (Other): Patients with AKI receive standard of care in the conventional manner by the primary clinicians
  Interventions: Other: Conventional management arm
- AKI sniffer instigated AKI management (Active Comparator): primary clinicians for the AKI patients in this arm receive a verbal alert and reminder of KDIGO guidelines.
  Interventions: Other: AKI sniffer instigated AKI management

INTERVENTIONS:
Other: Conventional management arm — Based on KDIGO guidelines and as per primary physician in the ICU
  Arms: Conventional management arm
Other: AKI sniffer instigated AKI management — After identification of patients with AKI by the sniffer, primary physicians will be notified about the development of the syndrome and will be given a copy of the KDIGO guidelines for management of AKI.
  Arms: AKI sniffer instigated AKI management

SUMMARY:
Introduction: Acute kidney injury (AKI) increases mortality, hospital cost, and rate of progression toward end stage kidney disease 1-4. Early diagnosis and management of AKI is known to improve the above mentioned outcomes.

Hypothesis: the investigators will design and validate an electronic surveillance tool to screen all the ICU admissions for the earlier, more efficient diagnosis of AKI and as a result improve the outcome of AKI in ICU patients.

Methods: the investigators plan to use the patient database, and AKIN (AKI network) definition to design an electronic alert system to allow clinicians discover patients who develop AKI. Then a randomized clinical trial will be conducted to compare earlier intervention (based on Kidney Disease: Improving Global Outcomes [KDIGO] guidelines) initiated by AKI sniffer alert to the conventional management provided by primary physician in ICU.

DETAILED DESCRIPTION:
A prospective controlled, unblinded clinical trial will be conducted among AKI patients who are detected by the use of AKI sniffer. The investigators will randomize consecutive patients who were detected to have AKI by AKI sniffer into two groups. In one group (control group), patients will receive standard clinical care by the primary ICU physicians. The primary physicians who take care of the control subjects will be kept blinded of the results of the AKI sniffer. All the ICU physicians will receive a copy of KDIGO (March 2012) guidelines for management of AKI prior to the initiation of the patient accrual. In the intervention group, the research team will inform the primary care team about the occurrence of the AKI and provides a copy of KDIGO guidelines for management of AKI to the clinicians. Each subject will be followed until hospital discharge or for a maximum of 3 months, for clinical and laboratory data including peak serum creatinine, creatinine at the end of follow up, peak AKIN stage, along with other secondary outcomes. The investigators will exclude the prevalent cases (AKI patients who have had AKI documented in their medical records by clinicians prior to the ICU admission).

ELIGIBILITY:
Inclusion Criteria:

* All patients who are admitted in adult ICUs in Mayo Clinic Rochester
* Foley catheter for hourly UOP measurement

Exclusion Criteria:

* Prisoners
* Patients less than 18 years old.
* Lack of research authorization (in control group)
* ESRD on dialysis or s/p kidney transplantation
* Known AKI before admission to ICU
* Moribund patients
* Prevalent AKI admission in ICU (patients who have diagnosis of AKI documented in their medical records prior to ICU admission)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2266 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
Change in acute kidney injury as measured by the Acute Kidney Injury Network Staging System | baseline, 4 weeks
  The Acute Kidney Injury Network staging system is based on data indicating that a small change in serum creatinine influences outcome. Increases in serum creatinine or decreased urine output indicate greater kidney injury, with the stage ranging from 1 to 3. The higher the number, the greater the kidney injury.

CONTACTS AND LOCATIONS:
Overall Officials: Kianoush Kashani, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
We plan to share IPD after initiation of patient recruitment.